CLINICAL TRIAL: NCT03532061
Title: Enhancing Family Caregivers' Strengths and Skills in Managing Older Cancer Patients
Brief Title: Caregivers' Strengths-Skills: Managing Older Cancer Patients' Symptoms
Acronym: FamCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 10-01719; 7R01CA115315-06 (NIH)
Record Dates: First submitted 2018-04-05; First posted 2018-05-22 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2019-05

CONDITIONS: Cancer
Keywords: Familial Caregiver; Cancer; Symptom Management; COPE Principles; Problem-solving Skills Training Program
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FamCare Group (Experimental): Family caregivers who receive 6 in-person problem-solving skills training sessions (FamCare Program).
  Interventions: Behavioral: FamCare Program
- Caregiver Support Group (Active Comparator): Family caregivers who receive 6 in-person caregiver support group sessions.
  Interventions: Other: Caregiver Support Group

INTERVENTIONS:
Behavioral: FamCare Program — 6 in-person sessions of biweekly home care problem-solving skills training (FamCare) delivered by a health educator.
  Arms: FamCare Group
Other: Caregiver Support Group — 6 in-person caregiver support group sessions held biweekly and moderated by a health educator.
  Arms: Caregiver Support Group

SUMMARY:
Caregiver education and training programs that specifically target caregiver informational and training needs during the survivorship period have been limited. In recognition of families' direct involvement in health care decision-making, health advocacy and care provision, programs are needed that can maximize families' caregiving abilities and skills and provide them with the information and resources they may need to identify and address elderly cancer patients' post-treatment symptom management. The goal of this study was to implement and evaluate the efficacy of a short-term problem-solving skills training program (relative to participating in a caregiver support group) for familial caregivers to lower income older (55+) post-treatment cancer patients.

DETAILED DESCRIPTION:
Cancer is one of the leading health disorders that can lead to impaired functioning and mortality in the elderly. With the aging of the population, more people will be living with a cancer diagnosis. The most dramatic increases will be among ethnic minorities. Advances in cancer detection and treatment are increasing cancer patients' survival and making it possible for many to be managed as outpatients and remain in the community. These advances have also contributed to an increased number of older adults living longer with/surviving for longer periods with having had cancer.

Recognition of the centrality of families' role in patients' treatment and recovery is widespread. Less attention, however, has been focused on developing programs and interventions that include or target the families' role during the cancer survivorship period, a period when patients are coping with the consequences of cancer and its treatment. During this period, when contact with the health care system is less intense, cancer patients' symptoms may go unrecognized or be poorly managed. Family members are directly involved in health care decision-making, functioning not only as a health care advocate for the elderly patient, but also ensuring that patients adhere to symptom management routines (e .g. encouraging them to take their pain medication, providing reassurance of the appropriateness of attending to certain symptoms). Family members' ongoing, frequent, contact with their elderly relative makes them ideally situated to monitor patients' functioning and detect subtle changes in their condition.

The goal of the proposed study was to implement and evaluate the utility of a brief training program to support and enhance the problem-solving caregiving skills of familial caregivers to facilitate optimum symptom control for older cancer patients during the post-treatment period. The rationale for this approach is based upon a diverse body of theoretical and empirical work. It represents a distillation and consolidation of research on cancer and the family, and draws from the broader bodies of work on disease management in the elderly, disparities in health care, cultural perspectives on illness, family caregiving in chronic disease, health behavior, health education and emerging approaches in palliative care.

Given the challenges patients and families may be experiencing during the post treatment period, ethical considerations mandated some type of service provision for the comparison condition. It was necessary to select an intervention that would be of potential benefit to the caregiver and/or the elderly patient, but would not necessarily be expected to directly impact the caregiver skills targeted in the Problem-solving condition. These considerations led to the selection of a caregiver support program as an acceptable comparison condition.

This investigation addresses a significant gap in the caregiver literature. While there is widespread recognition of the centrality of the family's role in long-term care situations, little attention has been focused on the post-treatment period. Programs that can empower familial caregivers and enhance their problem-solving strengths may enable them to be more effective in managing their relatives' care needs.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Have a cancer diagnosis
2. Have completed active treatment
3. Be an older adult, aged 55 or older
4. Have a family member who is their caregiver
5. Understand English or Spanish
6. Not be severely cognitively impaired

Patient Exclusion Criteria:

* Patient must be in the post-treatment period

Familial Caregiver Inclusion Criteria:

1. Be 18 or older
2. Live with or have frequent (at least weekly face-to-face) contact with patient
3. Understand English or Spanish

Familial Caregiver Exclusion Criteria:

* Not be severely cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-08-07 (Actual); Primary Completion 2011-04-14 (Actual); Study Completion 2011-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver Social Problem-Solving Inventory Scale Score | Baseline, 1 & 7 months post-intervention delivery
  Social Problem-Solving Inventory-Revised (SPSI-R:L): This is a 52 item instrument that measures one's ability to resolve problems encountered in everyday living. Scoring results in five standardized scale scores (1. Positive problem orientation; 2. Negative problem orientation; 3. Impulsivity/carelessness style; 4. Avoidance style; and 5. Rational problem solving), four Rational Problem Solving subscale scores (1. Problem definition formulation; 2. Generation of alternative solutions; 3. Decision making; and 4. Solution implementation and verification) and a Total SPSI-R:L standard score. Raw scores are converted to standard scores. The total SPSI-R:L score and each scale/subscale score has a mean of 100 and a standard deviation of 15. With the total SPSI-R:L score, higher scores indicate "good" social problem-solving ability. The extent to which "good" and "poor" problem-solving ability is demonstrated, is determined by observing how far the scores are from the mean score of 100.

SECONDARY OUTCOMES:
Caregiver's Satisfaction with Quality of Patient Care - FAMCARE Scale Score | Baseline, 1 & 7 months post-intervention delivery
  The impact of the short-term problem-solving skills training program on the caregiver's perceptions of and satisfaction with the quality of the patient's care relative to participating in the support condition, will be assessed utilizing the FAMCARE Scale. The FAMCARE Scale is a 20 item measure used to assess family satisfaction with health care of patients with advanced cancer. The scale contains 20 items and each item is a five-point Likert scale ranging from 1 (very satisfied) to 5 (very dissatisfied). The summary scale and individual subscales (Information giving, Availability of care, Physical care, and Pain control) are scored to range from 20-100, with high scores indicative of treatment/care dissatisfaction. To make the FAMCARE Scale easier to interpret, the scores were computed to reverse the scale such that higher values indicate higher satisfaction with care.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria H. Raveis, PhD, Principal Investigator — New York University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raveis VH, Tobin J, Karus D, Zhou R, Faber KE, Carrero M, Estrada I. Family caregiving to older, minority cancer survivors living in the community: Perspectives from a randomized control trial of caregiver problem-solving skills training. The Gerontologist 51(S2):496, 2011.
- [Background] Raveis VH, Tobin J, Karus D, Faber K, Zhou R, Carrero M, Estrada I. Family caregiving transitions: Addressing the care needs of older adults during the cancer survivorship period. The Gerontologist 50(S1): 475, 2010.
- [Result] Raveis VH, Karus D, Zhou R, Carrero-Tagle M, Faber K, Estrada I, Tobin JN. FamCare: Cognitive-behavioral problem solving training for family caregivers to cancer survivors. Gerontologist 56(Suppl_3): 684, 2016.